CLINICAL TRIAL: NCT05500313
Title: The Effect of Education and Counseling Based on HypnoBreastfeeding Philosophy on Breastfeeding Status, Breastfeeding Self-Efficacy and Breastfeeding Motivation
Brief Title: The Effect of Education and Counseling Based on HypnoBreastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, Associate Prof, Mersin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NS
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Hypno-breastfeeding Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypno-breastfeeding Education (Experimental): An announcement was made on social media platforms for hypno-breastfeeding education programme, and they were invited to the education. Pre-applicant women were informed about the education and research process and their informed consent was signed via e-mail. An average of 4-5 women were included in each group. this group, the training consisted of 4 sessions and a total of 12 hours. It included information about breastfeeding, hypnosis approaches and different techniques. In line with the demands of the group, the session days and hours were decided with together. The Hypno-Breastfeeding Education Programme was offered to each group in a maximum of 2 weeks.
  Interventions: Behavioral: Hypno-breastfeeding Education
- Standart Breastfeeding Education (Experimental): An announcement was made on social media platforms for standart breatfeeding education programme, and they were invited to the education. Pre-applicant women were informed about the education and research process and their informed consent was signed via e-mail.This education was done in one go. In this group, the training consisted of 1 sessions and a total of 3 hours. It included only information about breastfeeding.
  Interventions: Behavioral: Experimental: Standart Breastfeeding Education

INTERVENTIONS:
Behavioral: Hypno-breastfeeding Education — The hypnobreastfeeding education program consists of 4 sessions and 12 hours. It includes information about breastfeeding, mental preparation for the breastfeeding experience, emotional studies, motivational practices, awareness and self-compassion practices.
  Arms: Hypno-breastfeeding Education
Behavioral: Experimental: Standart Breastfeeding Education — The standard breastfeeding education program consists of 1 session and 3 hours. It contains only information and applications about breastfeeding.
  Arms: Standart Breastfeeding Education

SUMMARY:
The aim of this study is to determine the effect of education and counseling based on the hypno-breastfeeding philosophy given in the antenatal period on only breastfeeding status, breastfeeding self-efficacy and breastfeeding motivation.

DETAILED DESCRIPTION:
This is a non-randomized experimental study. Data were collected from 80 women who attended hypno-breastfeeding-based education or standart breastfeeding education from Turkey between September 2021 and February 2022. Participants who met the inclusion criteria were informed about the purpose of the study and hypno-breastfeeding-based education or standart breastfeeding education, informed consent was obtained from those who agreed to participate. Data were collected at the time of consent to the study, pre-education, post-education, 1 week and 8 weeks after birth. Collected by the first author. The CONSORT directive was followed in the planning, implementation and writing of the research.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to a healthy pregnancy,
* Native language is Turkish,
* Have single fetus
* Must be able to breastfeeding with her baby
* Must be able to join wit education.

Exclusion Criteria:

* Complications,
* Psychological or psychiatric disorder,
* Un-available follow-upps

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Level of breastfeeding self-efficacy | Between 28-34 weeks of pregnancy
  Women's breastfeeding self-efficacy during pregnancy were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al (2003) for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. (2010). This scale consisting of 14 items is a 5-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding self-efficacy | Between 30-36 weeks of pregnancy
  Women's breastfeeding self-efficacy during pregnancy were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al (2003) for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. (2010). This scale consisting of 14 items is a 5-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding self-efficacy | Postpartum 1st week
  Women's breastfeeding self-efficacy at the postpartum period were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al (2003) for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. (2010). This scale consisting of 14 items is a 5-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding motivation | Postpartum 1st week
  In order to improve the breastfeeding motivation of women in the postpartum period, Peleg et al. Breastfeeding Motivation Scale was developed by in 2015. The scale consists of 24 items and 5 sub-dimensions. The scale does not have a total score. The scores of the sub-dimensions are calculated by taking the average of the sub-dimension scores of the scale. As the score obtained from the scale sub-dimension increases, the motivation score representing that sub-dimension also increases. The Turkish adaptation of the scale was carried out by Mızrak and Özdoğan in 2017, and the cronbach alpha value was determined as 0.88.
Breastfeeding Process Evaluation Form | Postpartum 1st week
  The breastfeeding process evaluation form was created by the researchers as a result of the literature review in order to determine the status of exclusive breastfeeding in the first eight weeks and the factors affecting it. Breastfeeding processes evaluation form consists of 20 questions.
Level of breastfeeding self-efficacy | Postpartum 8 st week
  Women's breastfeeding self-efficacy at the postpartum period were evaluated with the Breastfeeding Self-efficacy Scale.
  This scale was developed by Dennis et al (2003) for fear after childbirth. The Turkish validity and reliability of the scale were performed by Tokat et al. (2010). This scale consisting of 14 items is a 5-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 14 to 70. The scale has no cutoff score, and high scores indicated higher breastfeedin self- efficacy.
  There are two versions of the scale used during pregnancy and postpartum. In both versions, the items are the same and the tenses change. In order to evaluate the Turkish validity and reliability of both antenatal and postnatal versions of the scale, language, structure and predictive validity analyzes were performed and the Cronbach's alpha value was found to be 0.87 for the antenatal measurement tool and 0.86 for the postnatal measurement tool.
Level of breastfeeding motivation | Postpartum 8 st week
  In order to improve the breastfeeding motivation of women in the postpartum period, Peleg et al. Breastfeeding Motivation Scale was developed by in 2015. The scale consists of 24 items and 5 sub-dimensions. The scale does not have a total score. The scores of the sub-dimensions are calculated by taking the average of the sub-dimension scores of the scale. As the score obtained from the scale sub-dimension increases, the motivation score representing that sub-dimension also increases. The Turkish adaptation of the scale was carried out by Mızrak and Özdoğan in 2017, and the cronbach alpha value was determined as 0.88.
Breastfeeding Process Evaluation Form | Postpartum 8 st week
  The breastfeeding process evaluation form was created by the researchers as a result of the literature review in order to determine the status of exclusive breastfeeding in the first eight weeks and the factors affecting it. Breastfeeding processes evaluation form consists of 20 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Gokce Isbir, Principal Investigator — Mersin University
Locations (1):
- Gozde Gokce Isbir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No